CLINICAL TRIAL: NCT06912607
Title: Balance and Fitness Enhancement Program for Deaf Older Adults
Brief Title: Exercise Program for Deaf Seniors to Increase Their Balance and Fitness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gallaudet University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY24-34; 1R15AG087454-01 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Deaf; Fall; American Sign Language; Old Age
Keywords: Exercise; Fall risk; Deaf; Senior citizen; Older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Group (Other): Deaf older adults.
  Interventions: Behavioral: Balance in Motion Exercise class

INTERVENTIONS:
Behavioral: Balance in Motion Exercise class — 8 weeks of 2 meetings/wk exercise class, with a once weekly homework exercise, delivered entirely in ASL

SUMMARY:
Deaf older adults 60 years and older are enrolled into an 8-week exercise program delivered in American Sign Language. The class meets twice a week, with handout and video homework.

Outcome measures are self-reported balance confidence, lower extremity strength, walking and agility, and standing balance. In addition, attendance and keeping up with exercises at home will be tracked.

DETAILED DESCRIPTION:
The intervention will be 8 weeks of 2 meetings/wk exercise class, delivered entirely in ASL.

Homework exercise will also be provided.

10-12 participants will be recruited for each of the 4 semesters of offerings.

Physical balance as well as balance confidence will be measured prior to and immediately after the 8-week intervention. In addition, balance confidence will be measured 6-months after the conclusion of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Deaf
* Uses American Sign Language (ASL) fluently
* Community-dwelling
* Able to walk independently for at least 20 ft
* Willing to attend classes twice a week at Gallaudet University

Exclusion Criteria:

* Blindness
* Dementia
* Neurological conditions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Sit-to-Stand | 1 - 21 days before the start of intervention; within 2 weeks of the end of intervention
  The number of times a person can stand from a chair and sit down, without using hands.
Timed Up-and-Go | 1 - 21 days before the start of intervention; within 2 weeks of the end of intervention
  The time it takes for a person to stand from a chair, walk 10 ft, turn around, walk back, and sit back down.
Modified Clinical Test of Sensory Integration on Balance | 1 - 21 days before the start of intervention; within 2 weeks of the end of intervention
  The measure of how steadily a person can stand under 4 conditions (eyes open, on firm surface, eyes closed on firm surface, eyes open on foam, and eyes closed on foam)
Sit and Reach | 1 - 21 days before the start of intervention; within 2 weeks of the end of intervention
  How far a person can reach beyond their toes. Measure of flexibility.
Activities-specific Balance Confidence scale | 1 - 21 days before the start of intervention; within 2 weeks of the end of intervention, 6 months after intervention
  A self-report measure of how confident a person is in not falling under various conditions. Reported in 0-100%; higher score means more confidence (better outcome).
Fall Risk Questionnaire | 1 - 21 days before the start of intervention; within 2 weeks of the end of intervention, 6 months after intervention
  A self-report measure of the number of risk factors a person exhibits. Reported in a scale of 0-14 points; higher score indicates a greater risk (worse outcome).

SECONDARY OUTCOMES:
Attendance rate | During intervention
  How many exercise class sessions, out of 16, a participant attended
Step Count | During intervention
  The number of steps gathered through Fitbit
Effective exercise level | During intervention
  The Active Zone Minutes gathered through Fitbit
Self-reported exercise level | 6 months after the intervention
  The participant's report on how much time they are spending on exercises

CONTACTS AND LOCATIONS:
Overall Officials: Chizuko Tamaki, AuD, PhD, Principal Investigator — Gallaudet University
Locations (1):
- Gallaudet University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided